CLINICAL TRIAL: NCT06417411
Title: A Prospective, Randomized Controlled Study to Evaluate the Effects of Daily Low Dose Aspirin in Pregnant Women With Sickle Cell Disease When Initiated at the First Trimester Versus the Second Trimester of the Gestational Period
Brief Title: LEARNER- Low dosE AspiRiN prEterm tRial (Angola)
Acronym: LEARNER
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Investigacao em Saude, Angola (Other Government)
Collaborators: FUNDACIÓN BANCARIA CAIXA D'ESTALVIS I PENSIONS DE BARCELONA (Unknown); FUNDAÇAO CALOUSTE GULBENKIAN (Unknown); CLINCOORD SERVICES, INC. (Unknown); CLINCOORD PRESTAÇÃO DE SEVIÇOS, LDA ANGOLA (Unknown); Escola Superior de Tecnologia da Saúde de Lisboa (Other); ClinCoord Research Center at Luanda Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LEARNER
Record Dates: First submitted 2024-05-02; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Sickle Cell Disease; Pregnancy Related; Pregnancy Complications; Pre-Eclampsia
Keywords: LEARNER; ANGOLA; Maternidade Lucrécia Paim; Hospital Materno Infantil Dr Manuel Pedro Azancot de Menezes; Aspirin; Capacity Building
MeSH Terms: conditions — Anemia, Sickle Cell; Pregnancy Complications; Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin in First trimester (Active Comparator): Participants who will start the study medication (Aspirin) during the first trimester
  Interventions: Drug: Aspirin 100mg
- Aspirin in Second trimester (Experimental): Participants who will start the study medication (Aspirin) during the second trimester
  Interventions: Drug: Aspirin 100mg

INTERVENTIONS:
Drug: Aspirin 100mg — Daily use of low dose aspirin.

SUMMARY:
This study is being conducted to evaluate the safety and effect of starting daily use of low dose (100 mg) aspirin in pregnant women with sickle cell disease, who are being followed in two county hospitals in Angola, in the first trimester versus the second trimester of the gestational period.

DETAILED DESCRIPTION:
The proposed project is a prospective, randomized controlled study to evaluate the effects of daily low dose aspirin in pregnant women with Sickle Cell Disease at the first trimester versus the second trimester of the gestation period.

The study will include 450 female participants of all ages, in multiple maternity hospitals in Luanda, Angola, with an official diagnosis of Sickle Cell Disease and confirmed pregnancy. Patients who consent to take part in the study will be given 100 mg aspirin once daily either at the first trimester (6-13 weeks) or the second trimester (14-27 weeks) of the gestation period. Up to 450 participants will be randomly assigned in a 1:1 ratio to the two study treatment trimester groups (225 starting the low dose of aspirin at the first trimester and 225 starting the low dose of aspirin at the second trimester). In both treatment arms, daily use of low dose aspirin will be prescribed/administered until week 36 or time of delivery, whichever comes earlier.

Study Duration:

Each participant will be enrolled in the study for the duration of the pregnancy as follow:

Screening Visit Randomized Treatment Period Follow Up Period (6 weeks postpartum)

ELIGIBILITY:
Inclusion Criteria:

* 1. Pregnant women with Sickle Cell Disease 15 years old and older
* 2. Attending Maternidade Lucrecia Paim, Hospital Materno Infantil Dr. Manuel Pedro Azancot de Menezes, or any health commodities in the neighboring area of the referred hospitals
* 3. Willing to attend the regular consultations, and consent to take part in the study.

Exclusion Criteria:

* 1. Pregnant women with Sickle Cell Disease in the third trimester (after week 27)
* 2. HIV infection
* 3. Diabetes mellitus
* 4. Chronic hypertension
* 5. Liver disease measured by laboratory indication being 3 times above the upper limit of normal
* 6. Sickle nephropathy
* 7. Multiple pregnancies
* 8. Hypersensitivity to aspirin
* 9. History of blood transfusion in the last 3 months
* 10.Those who did not consent to participate in the study.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 450 (Estimated)
Dates: Start 2024-03-16 (Actual); Primary Completion 2025-03-16 (Estimated); Study Completion 2026-03-16 (Estimated)

PRIMARY OUTCOMES:
Maternal Mortality | 2 years
  Measuring the number of maternal mortalities up to 6 weeks postpartum.
Life Birth Related Events | 2 years
  The number of preterm births will be measured by the number of deliveries before 37 weeks gestational age.
Late Abortion Related Events | 2 years
  Measuring the number of unintentional abortions late in the pregnancy

SECONDARY OUTCOMES:
Maternal Morbidity | 2 years
  hypertensive disorders, vaginal bleeding, antepartum hemorrhage, and postpartum hemorrhage, will be aggregated to determine the number of morbidity events related to the mother.
Fetal Mortality Outcomes | 2 years
  fetal loss due to small gestational age, perinatal mortality, spontaneous abortion, and stillbirth, will be aggregated to quantify the number of fetal mortality events.
Other Fetal Events | 2 years
  Early preterm delivery (less than 34 weeks of gestation), extreme preterm delivery (less than 28 weeks of gestation), actual birth weight (measured in grams), post-term delivery (more than 42 weeks of gestation) will be combined to report the number of other fetal related events.

OTHER OUTCOMES:
Clinical Research Personnel Capacity Building | 2 years
  The number of investigators and research staff successfully trained will be combined to measure the ability of conducting clinical research and data capture by otherwise research naive personnel.
Institutional Collaborations | 2 years
  The number of institutions involved in the conduction of the LEARNER project will be reported to measure collaboration between Angolan scientific/medical institutions and other international research entities.

CONTACTS AND LOCATIONS:
Overall Officials: JOANA MORAIS, PhD, Principal Investigator — INSTITUTO NACIONAL DE INVESTIGAÇÃO EM SAÚDE; TATIANA GOMES, BA/BS/Pre-MD, Study Director — ClinCoord
Locations (1):
- Instituto Nacional de Investigação Em Saúde, Luanda, Angola

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borges E, Tchonhi C, Couto CSB, Gomes V, Amorim A, Prata MJ, Brito M. Unusual beta-Globin Haplotype Distribution in Newborns from Bengo, Angola. Hemoglobin. 2019 May;43(3):149-154. doi: 10.1080/03630269.2019.1647230. Epub 2019 Aug 8. PMID 31394941
- [Background] Afolabi BB, Babah OA, Adeyemo TA, Odukoya OO, Ezeaka CV, Nwaiwu O, Oshodi YA, Ogunnaike BA. Low-dose aspirin for preventing intrauterine growth restriction and pre-eclampsia in sickle cell pregnancy (PIPSICKLE): a randomised controlled trial (study protocol). BMJ Open. 2021 Aug 13;11(8):e047949. doi: 10.1136/bmjopen-2020-047949. PMID 34389570
- [Background] Atallah A, Lecarpentier E, Goffinet F, Doret-Dion M, Gaucherand P, Tsatsaris V. Aspirin for Prevention of Preeclampsia. Drugs. 2017 Nov;77(17):1819-1831. doi: 10.1007/s40265-017-0823-0. PMID 29039130